CLINICAL TRIAL: NCT03994224
Title: A Prospective Longitudinal Study of Fecal Microbiome and Calprotectin to Predict Response to Biological Therapy in Patients With Crohn's Disease
Brief Title: A Prospective Longitudinal Study of Fecal Microbiome and Calprotectin to Predict Response to Biological Therapy in Patients With CD
Status: Terminated | Type: Observational
Why Stopped: Decision made by team of investigators
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Siew Chien NG, Profressor, Chinese University of Hong Kong
Other Study IDs: CD MiRES
Record Dates: First submitted 2019-06-20; First posted 2019-06-21 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: Crohn Disease; Perianal Crohn Disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Crohn's disease (CD) is a chronic relapsing-remitting systemic inflammatory disease, affecting any part of the gastrointestinal tract. Biological therapy with anti-tumor necrosis factor (TNF) alpha is the established treatment of choice for the management of moderate to severe Crohn's disease. However, its efficacy in an individual patient is the unpredictable and long-term outcome is still suboptimal. Identifying biomarkers which can predict treatment response is thus of utmost importance and can allow personalized management.

In inflammatory bowel disease (IBD), altered fecal microbiota signatures have been consistently reported. Moreover, overall bacterial diversity is consistently decreased during intestinal inflammation.

Fecal calprotectin (FC) is a calcium and zinc binding protein largely confined to the neutrophil granulocytes and macrophages and is a very sensitive marker for detection of inflammation in the gastrointestinal tract.

C reactive protein (CRP) is an acute phase reactant. CD Patients with elevated baseline CRP levels responded to infliximab treatment better and early normalisation of CRP correlated with sustained long-term response to infliximab therapy.

The investigators hypothesize that faecal microbial signatures in conjunction with faecal calprotectin and CRP may have a role in predicting response to biological therapy in CD patients.

DETAILED DESCRIPTION:
Crohn's disease (CD) is a chronic relapsing-remitting systemic inflammatory disease, affecting any part of the gastrointestinal tract. Patients frequently present with abdominal pain, fever, and symptoms of bowel obstruction or diarrhea with passage of blood or mucus, or both. It can lead to significant morbidity and disability in some cases. Population-based studies revealed that up to 50% of CD patients required surgery within 10 years from diagnosis.Only 24% remain in remission over their lifetime disease course.

Biological therapy with anti-tumor necrosis factor (TNF) alpha is the established treatment of choice for the management of moderate to severe Crohn's disease. However, its efficacy in an individual patient is the unpredictable and long-term outcome is still suboptimal. Almost one-third of CD patients showed no response to anti-TNF and two-thirds do not achieve remission.The rate of loss of response after 1 year of infliximab therapy ranges between 23% and 46%.4 Identifying biomarkers which can predict treatment response is thus of utmost importance and can allow personalized management.

Several biomarkers have been identified in predicting treatment response. C reactive protein (CRP) is an acute phase reactant with a short half-life of only 19 hours. CD Patients with elevated baseline CRP levels (>3mg/L) responded to infliximab treatment better and early normalisation of CRP correlated with sustained long-term response to infliximab therapy. Similar results were shown in adalimumab therapy. CD patients who had achieved normalisation of CRP (<3mg/L) at both week 4 and week 12 were less likely to discontinue adalimumab and had sustained clinical benefit.

Fecal calprotectin (FC) is a calcium and zinc binding protein largely confined to the neutrophil granulocytes and macrophages and is a very sensitive marker for detection of inflammation in the gastrointestinal tract. FC levels dropped significantly in CD patients who responded to infliximab therapy. A decrease in FC level after therapy has been demonstrated to be associated with clinical, endoscopic and histological improvements. Moreover, a study has demonstrated that combination of CRP and FC represented a good predictor of relapse of CD among patients on anti-metabolite therapy after infliximab was stopped.

In inflammatory bowel disease , altered fecal microbiota signatures have been consistently reported which included a reduction in biodiversity with lower proportions of Firmicutes and increases in Proteobacteria and Bacteroidetes phylum members.Moreover, overall bacterial diversity is consistently decreased during intestinal inflammation. Besides, CD patients have richer fungal species and higher microbiome diversities in mucosal biopsies. Several fungal species, including Candida spp., Gibberella moniliformis, Alternaria brassicicola and Cryptococcus neoformans, are increased in tissues from CD patients. CD patients may harbor increased numbers of bacteriophages in inflamed tissue and feces, though no specific viruses have been associated with human IBDs to date.

Few studies have studied the longitudinal changes in the gut microbiome with drug treatment in IBD. Shaw et al. characterized 19 children with CD and 4 with ulcerative colitis (UC), showing that dysbiosis at baseline correlated with the degree of inflammatory burden of luminal disease. An improvement in fecal diversity was seen with clinical response in UC but not CD.Restoration of gut diversity has been reported previously with anti-TNF therapy. However, a more diverse microbiome has not been previously shown to be predictive of treatment response in children. Recent study by the Massachusetts group including 85 IBD patients (43 UC, 42 CD) who initiated treatment with vedolizumab revealed that baseline microbiome was significantly higher and Roseburia inulinivorans and a Burkholderiales species were more abundant at baseline among CD patients achieving week 14 remission. Patients achieving remission at week 14 demonstrated persistency in the microbial composition at both week 30 and week 54, suggesting that attainment of remission at week 14 is associated with durable changes in microbiomes. Thus, early changes in microbiome could help identify patients who will likely to achieve and maintain response to treatment.

The investigators hypothesize that faecal microbial signatures in conjunction with faecal calprotectin and CRP may have a role in predicting response to biological therapy in CD patients.

ELIGIBILITY:
Inclusion Criteria:

Patients with moderate to severe Crohn's disease

1. Aged ≥ 18 years old
2. Confirmed diagnosis of Crohn's disease according to established clinical, endoscopic and histological criteria
3. Moderate to severe Crohn's disease who are due to start biological therapy
4. Written informed consent obtained

Subjects with perianal Crohn's disease

1. Aged ≥ 18 years old
2. Confirmed diagnosis of Crohn's disease with perianal involvement according to established clinical, endoscopic and histological criteria
3. Subjects with active perianal Crohn's disease who are due to start biological therapy
4. Written informed consent obtained

4.2. Exclusion Criteria

1. Previous bowel surgery/ stoma
2. History of anti-TNF use in the last 3 months
3. Malignant disease within 5 years
4. Use of probiotics, prebiotics or antibiotics in the past 1 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive CD subjects who visit Prince of Wales Hospital in Hong Kong
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2019-02-18 (Actual); Primary Completion 2022-08-29 (Actual); Study Completion 2022-08-29 (Actual)

PRIMARY OUTCOMES:
Asymptomatic Crohn's Disease patients | 2 years
  Defined as normal CRP level <10mg/l and no use of corticosteroid in the last 4 weeks.
Asymptomatic perianal Crohn's Disease patients | 2 years
  Defined as the absence of draining fistula on two consecutive visits according to Fistula Drainage Assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Siew Chien Ng, Prof, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Hong Kong, Hong Kong

REFERENCES:
- [Background] Aniwan S, Park SH, Loftus EV Jr. Epidemiology, Natural History, and Risk Stratification of Crohn's Disease. Gastroenterol Clin North Am. 2017 Sep;46(3):463-480. doi: 10.1016/j.gtc.2017.05.003. Epub 2017 Jul 19. PMID 28838409
- [Background] Silverstein MD, Loftus EV, Sandborn WJ, Tremaine WJ, Feagan BG, Nietert PJ, Harmsen WS, Zinsmeister AR. Clinical course and costs of care for Crohn's disease: Markov model analysis of a population-based cohort. Gastroenterology. 1999 Jul;117(1):49-57. doi: 10.1016/s0016-5085(99)70549-4. PMID 10381909
- [Background] Allez M, Karmiris K, Louis E, Van Assche G, Ben-Horin S, Klein A, Van der Woude J, Baert F, Eliakim R, Katsanos K, Brynskov J, Steinwurz F, Danese S, Vermeire S, Teillaud JL, Lemann M, Chowers Y. Report of the ECCO pathogenesis workshop on anti-TNF therapy failures in inflammatory bowel diseases: definitions, frequency and pharmacological aspects. J Crohns Colitis. 2010 Oct;4(4):355-66. doi: 10.1016/j.crohns.2010.04.004. Epub 2010 Jun 29. PMID 21122530
- [Background] Billiet T, Cleynen I, Ballet V, Ferrante M, Van Assche G, Gils A, Vermeire S. Prognostic factors for long-term infliximab treatment in Crohn's disease patients: a 20-year single centre experience. Aliment Pharmacol Ther. 2016 Oct;44(7):673-83. doi: 10.1111/apt.13754. Epub 2016 Aug 9. PMID 27502581
- [Background] Reinisch W, Wang Y, Oddens BJ, Link R. C-reactive protein, an indicator for maintained response or remission to infliximab in patients with Crohn's disease: a post-hoc analysis from ACCENT I. Aliment Pharmacol Ther. 2012 Mar;35(5):568-76. doi: 10.1111/j.1365-2036.2011.04987.x. Epub 2012 Jan 18. PMID 22251435
- [Background] Jurgens M, Mahachie John JM, Cleynen I, Schnitzler F, Fidder H, van Moerkercke W, Ballet V, Noman M, Hoffman I, van Assche G, Rutgeerts PJ, van Steen K, Vermeire S. Levels of C-reactive protein are associated with response to infliximab therapy in patients with Crohn's disease. Clin Gastroenterol Hepatol. 2011 May;9(5):421-7.e1. doi: 10.1016/j.cgh.2011.02.008. Epub 2011 Feb 17. PMID 21334460
- [Background] Karmiris K, Paintaud G, Noman M, Magdelaine-Beuzelin C, Ferrante M, Degenne D, Claes K, Coopman T, Van Schuerbeek N, Van Assche G, Vermeire S, Rutgeerts P. Influence of trough serum levels and immunogenicity on long-term outcome of adalimumab therapy in Crohn's disease. Gastroenterology. 2009 Nov;137(5):1628-40. doi: 10.1053/j.gastro.2009.07.062. Epub 2009 Aug 5. PMID 19664627
- [Background] Kiss LS, Szamosi T, Molnar T, Miheller P, Lakatos L, Vincze A, Palatka K, Barta Z, Gasztonyi B, Salamon A, Horvath G, Toth GT, Farkas K, Banai J, Tulassay Z, Nagy F, Szenes M, Veres G, Lovasz BD, Vegh Z, Golovics PA, Szathmari M, Papp M, Lakatos PL; Hungarian IBD Study Group. Early clinical remission and normalisation of CRP are the strongest predictors of efficacy, mucosal healing and dose escalation during the first year of adalimumab therapy in Crohn's disease. Aliment Pharmacol Ther. 2011 Oct;34(8):911-22. doi: 10.1111/j.1365-2036.2011.04827.x. Epub 2011 Aug 24. PMID 21883326
- [Background] Boschetti G, Garnero P, Moussata D, Cuerq C, Preaudat C, Duclaux-Loras R, Mialon A, Drai J, Flourie B, Nancey S. Accuracies of serum and fecal S100 proteins (calprotectin and calgranulin C) to predict the response to TNF antagonists in patients with Crohn's disease. Inflamm Bowel Dis. 2015 Feb;21(2):331-6. doi: 10.1097/MIB.0000000000000273. PMID 25625487
- [Background] Guidi L, Marzo M, Andrisani G, Felice C, Pugliese D, Mocci G, Nardone O, De Vitis I, Papa A, Rapaccini G, Forni F, Armuzzi A. Faecal calprotectin assay after induction with anti-Tumour Necrosis Factor alpha agents in inflammatory bowel disease: Prediction of clinical response and mucosal healing at one year. Dig Liver Dis. 2014 Nov;46(11):974-9. doi: 10.1016/j.dld.2014.07.013. Epub 2014 Aug 2. PMID 25096964
- [Background] Roseth AG, Aadland E, Grzyb K. Normalization of faecal calprotectin: a predictor of mucosal healing in patients with inflammatory bowel disease. Scand J Gastroenterol. 2004 Oct;39(10):1017-20. doi: 10.1080/00365520410007971. No abstract available. PMID 15513345
- [Background] Sipponen T, Savilahti E, Karkkainen P, Kolho KL, Nuutinen H, Turunen U, Farkkila M. Fecal calprotectin, lactoferrin, and endoscopic disease activity in monitoring anti-TNF-alpha therapy for Crohn's disease. Inflamm Bowel Dis. 2008 Oct;14(10):1392-8. doi: 10.1002/ibd.20490. PMID 18484671
- [Background] Louis E, Mary JY, Vernier-Massouille G, Grimaud JC, Bouhnik Y, Laharie D, Dupas JL, Pillant H, Picon L, Veyrac M, Flamant M, Savoye G, Jian R, Devos M, Porcher R, Paintaud G, Piver E, Colombel JF, Lemann M; Groupe D'etudes Therapeutiques Des Affections Inflammatoires Digestives. Maintenance of remission among patients with Crohn's disease on antimetabolite therapy after infliximab therapy is stopped. Gastroenterology. 2012 Jan;142(1):63-70.e5; quiz e31. doi: 10.1053/j.gastro.2011.09.034. Epub 2011 Sep 22. PMID 21945953
- [Background] Sartor RB, Wu GD. Roles for Intestinal Bacteria, Viruses, and Fungi in Pathogenesis of Inflammatory Bowel Diseases and Therapeutic Approaches. Gastroenterology. 2017 Feb;152(2):327-339.e4. doi: 10.1053/j.gastro.2016.10.012. Epub 2016 Oct 18. PMID 27769810
- [Background] Hansen JJ, Sartor RB. Therapeutic Manipulation of the Microbiome in IBD: Current Results and Future Approaches. Curr Treat Options Gastroenterol. 2015 Mar;13(1):105-20. doi: 10.1007/s11938-014-0042-7. PMID 25595930
- [Background] Perez-Brocal V, Garcia-Lopez R, Vazquez-Castellanos JF, Nos P, Beltran B, Latorre A, Moya A. Study of the viral and microbial communities associated with Crohn's disease: a metagenomic approach. Clin Transl Gastroenterol. 2013 Jun 13;4(6):e36. doi: 10.1038/ctg.2013.9. PMID 23760301
- [Background] Wagner J, Maksimovic J, Farries G, Sim WH, Bishop RF, Cameron DJ, Catto-Smith AG, Kirkwood CD. Bacteriophages in gut samples from pediatric Crohn's disease patients: metagenomic analysis using 454 pyrosequencing. Inflamm Bowel Dis. 2013 Jul;19(8):1598-608. doi: 10.1097/MIB.0b013e318292477c. PMID 23749273
- [Background] Shaw KA, Bertha M, Hofmekler T, Chopra P, Vatanen T, Srivatsa A, Prince J, Kumar A, Sauer C, Zwick ME, Satten GA, Kostic AD, Mulle JG, Xavier RJ, Kugathasan S. Dysbiosis, inflammation, and response to treatment: a longitudinal study of pediatric subjects with newly diagnosed inflammatory bowel disease. Genome Med. 2016 Jul 13;8(1):75. doi: 10.1186/s13073-016-0331-y. PMID 27412252
- [Background] Lewis JD, Chen EZ, Baldassano RN, Otley AR, Griffiths AM, Lee D, Bittinger K, Bailey A, Friedman ES, Hoffmann C, Albenberg L, Sinha R, Compher C, Gilroy E, Nessel L, Grant A, Chehoud C, Li H, Wu GD, Bushman FD. Inflammation, Antibiotics, and Diet as Environmental Stressors of the Gut Microbiome in Pediatric Crohn's Disease. Cell Host Microbe. 2015 Oct 14;18(4):489-500. doi: 10.1016/j.chom.2015.09.008. PMID 26468751
- [Background] Ananthakrishnan AN, Luo C, Yajnik V, Khalili H, Garber JJ, Stevens BW, Cleland T, Xavier RJ. Gut Microbiome Function Predicts Response to Anti-integrin Biologic Therapy in Inflammatory Bowel Diseases. Cell Host Microbe. 2017 May 10;21(5):603-610.e3. doi: 10.1016/j.chom.2017.04.010. PMID 28494241